

# **PROTOCOL**

# **EGERS**

**European Geriatric Emergency Departments Registry Study** 

On Behalf of the Geriatrics EuSEM Interest Group and the EUSEM Research committee

Protocol Number: .....

Status: Version 2.3

Date: 20/09/2020



| STUDY PROTOCOL | |
|---|---|
| PROTOCOL NUMBER: | |
| TITEL: | |
| The European Geriatric Emergency Departments Registry Study | |
| PROMOTER: | |
| European Society of Emergency Medicine (EuSEM). The EuSEM office is located at: Antwerpsesteenweg 124 B27 B-2630 Aartselaar, Brussels Belgium | |
| STUDY COORDINATORS: | |
| Principal Investigator: Assoc Prof Dr Mehmet Akif KARAMERCAN, Gazi University Faculty Medicine Emergency Medicine Department, Ankara/TURKEY (EuSEM Research Committe Member) | |
| Co-Principal Investigator: Assoc Prof Dr Zerrin Defne DÜNDAR, Konya/TURKEY (EuSE Research Committee Member) | EΜ |
| EGERS Steering Committee: | |
| Chair: Mehmet Akif KARAMERCAN (Turkey)<br>Co-Chair: Zerrin Defne DÜNDAR (Turkey) | |

### AND COUNTRY PI of THE STUDY

TECHNICAL SECRETARY:

**EuSEM Research Committee** 



#### 1. SUMARY

#### 1. STUDY PROMOTER

European Society of Emergency Medicine (EuSEM). The EuSEM office is located at:
Antwerpsesteenweg 124 B27
B-2630 Aartselaar, Brussels
Belgium

#### 2. STUDY TITEL

The European Geriatric Emergency Departments Registry Study (EGERS Study)

# 3. STUDY CODE EuSEM .....

#### 4. RESEARCHERS

Physicians of each participating center.

#### 5. PARTICIPATING CENTRES

European Emergency Departments (EDs)

#### 6. EVALUTED BY ETHICAL COMMITTEE

Local Ethical Committees.

#### 7. MONITOR RESPONSABLE

Non applicable.

#### 8. TREATMENT

Non applicable.

#### 9. PHASE OF STUDY

Non applicable.



#### 10. STUDY OBJETIVE

Principle Objective: Description of Epidemiologic and Age Related Characteristic of geriatric patients presenting to the ED

Secondary Objective: Determination of the prognostic and predictive values of vital sign based triage scores (REMS, MEWS and VIEWS Scores) regarding hospitalization, ICU admission and in-hospital mortality for geriatric patients presenting to ED

#### 11. DESIGN

Prospective multicentre observational study.

#### 12. DISEASES OF INTEREST

Non applicable.

#### 13. OUTCOME VARIABLE

Length of stay in the ED and Length of stay in the hospital if hospitalized. Status at 30 days: alive or dead.

#### 14. STUDY POPULATION AND SAMPLE SIZE

Patients  $\geq$  65 years of age those presented to EDs with any symptom Sample is generated with consecutive patients attending to EDs during study period.

#### 15. STUDY PERIOD

From 19th October 2020 to 16<sup>th</sup> November 2020, seven consecutive days of recruitment.



#### 2. GENERAL INFORMATION

A. Study Identification

| 1. Study Code Eus | SEM |
|---|---|
| Title: The European Ger. (EGERS Study). | iatric Emergency Departments Registry Study |
| B. Study Design | |
| Observational study | |
| C. Study final products | |
| Non applicable. | |
| D. <u>Promoter</u> | |
| European Society of Eme<br>The EuSEM office is loca<br>Antwerpsesteenweg 124<br>B-2630 Aartselaar, Bruss<br>Belgium | B27 |
| E. <u>Biological samples res</u> | <u>ponsible</u> |
| Non applicable. | |
| F. <u>Study monitors</u> | |
| Non applicable. | |
| G. Researchers and Cente | ers (recruitment still ongoing) |
| For countries represented of the RN. | in the EUSEM Research network, the country PI is the country Lead |



#### 3. INTRODUCTION, HYPOTHESIS AND OBJECTIVES

#### 3.1 Background

risen. The number of adults over 65 years of age who are presenting to emergency services is increasing in parallel with the prolongation of the average life expectancy (1). While geriatric presentations to emergency services comprise 40-50% of all emergency service presentations in the U.S., it has been reported that 3–23% of all emergency service presentations from various regions of the country comprise patients of 65 years of age and older (2-4). There are specific management practices for patients who are 65 years and older at emergency services due to the presence of comorbidities and the change of physiological responses to acute diseases in advanced age (1,2). Several risk-scoring systems have been developed to define the severity class of the patient during their initial evaluation at emergency services and generally named as Early Warning Scores (5–6). Early Warning Scores (EWS) incorporate physiological measurements, which do predict outcome although the addition of other simple clinical parameters might further improve the sensitivity and specificity of these scores (7). On the other hand all these EWS are simple and easy to calculate, making their use appropriate in an emergency setting (7). Of these EWS, the Modified Early Warning Score (MEWS), and the Rapid Emergency Medicine Score (REMS) have been widely used for many years (8) and The Vital PAC Early Warning Score (VIEWS) score was recently developed for the same purpose (9, 10).

Due to improved prevention, diagnosis and treatment modalities, life expectancy worldwide has

Only a few studies in the literature have evaluated risk-scoring systems for the geriatric patient group. Several studies have reported that risk-scoring systems, such as Identification of Seniors at Risk (ISAR) and Triage Risk Screening Tool (TRST), which are specifically developed for geriatric patients over 65 years who present to emergency services, are not sufficiently effective for evaluating



patients in more severe conditions (11,12). Other studies have reported that the ESI triage classification predicts the prognosis correctly in only half of the patients over 65 years of age (7,13). In another study that evaluated the MEWS for the geriatric patient group, which was calculated during the presentation in emergency services, has been stated to have a prognostic value in terms of a poor result (14).

Previously the TEDGeS (Turkish Emergency Departments Geriatric Scoring Study) pilot study was carried out and published (15,16). This study enrolled all geriatric patients (age  $\geq$  65 years) and carried out in 13 centers (University Hospitals, Government Education and Research Hospitals and Military Hospital ED) from different cities of Turkey.

#### **Key findings were:**

- Overall 30 % of hospitalized patients from ED are elderly patients and 30 % of these hospitalized patients were ICU hospitalizations
- In hospital mortality rate is about 6 % which is very high for general hospitalized patients
- The most common presenting symptoms are related to gastrointestinal systems and about 80
   % of the cases using at least one chronic medication (22.2 % of the cases using more than 4 chronic medications
- About 45 % of the cases final diagnosis are related to cardiovascular system and gastrointestinal system and nearly 85 % of the hospitalized cases are treated in non-surgical clinics (cardiology-pulmonology-internal medicine 65 %)
- MEWS, VIEWS and REMS scores are significantly high in hospitalized patients compared to discharged from ED and also these three scores are high in ICU hospitalized patients compared to both ward hospitalized and discharged patients.



- MEWS, VIEWS and REMS scores are significantly high in non-survivors compared to survivors
- MEWS, VIEWS scores has higher sensitivity and specificity in terms of in-hospital mortality

These results suggest that geriatric patients not only constitute significant proportion of ED presentations but also they need more hospitalization. The predictive powers of the MEWS, VIEWS and REMS scores for hospitalization and mortality in geriatric patients those presented to ED are significantly high and might be concerned in the ED triage of these patients.

#### References

- 1. Pines JM, Mullins PM, Cooper JK, Feng LB, Roth KE. National trends in emergency department use, care patterns, and quality of care of older adults in the United States. J Am Geriatr Soc 2013;61:12-7.
- 2. Roberts DC, McKay MP, Shaffer A. Increasing rates of emergency department visits for elderly patients in the United States, 1993 to 2003. Ann Emerg Med 2008;51:769-74.
- 3. Baz U, Satar S, Kozaci N, Acikalin A, Gulen M, Karakurt U. Geriatric patient admissions to emergency service. JAEM 2013, in press
- 4. Kekec Z, Koc F, Buyuk S. Review of geriatric patients hospitalization in emergency department. JAEM 2009;8(3):21-4.



- 5. Platts-Mills TF, Travers D, Biese K, et al. Accuracy of the Emergency Severity Index triage instrument for identifying elder emergency department patients receiving an immediate life-saving intervention. Acad Emerg Med 2010;17:238-43.
- 6. Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJ Med 2001;94:521-6.
- 7. Wheeler I, Price C, Sitch A, Banda P, Kellett J, Nyirenda M, Rylance J. Early warning scores generated in developed healthcare settings are not sufficient at predicting early mortality in Blantyre, Malawi: a prospective cohort study. PLoS One 2013;8(3): e59830.
- Olsson T, Terent A, Lind L. Rapid Emergency Medicine Score: a new prognostic tool for inhospital mortality in nonsurgical emergency department patients. J Intern Med 2004;255:579-87.
- 9. Prytherch DR, Smith GB, Schmidt PE, Featherstone PI. ViEWS--Towards a national early warning score for detecting adult inpatient deterioration. Resuscitation 2010;81:932-7.
- 10. Bleyer AJ, Vidya S, Russell GB, et al. Longitudinal analysis of one million vital signs in patients in an academic medical center. Resuscitation 2011;82:1387-92.
- 11. Salvi F, Morichi V, Grilli A, et al. Predictive validity of the Identification of Seniors At Risk (ISAR) screening tool in elderly patients presenting to two Italian Emergency Departments.
  Aging Clin Exp Res 2009;21:69-75.
- 12. Buurman BM, van den Berg W, Korevaar JC, Milisen K, de Haan RJ, de Rooij SE. Risk for poor outcomes in older patients discharged from an emergency department: feasibility of four screening instruments. Eur J Emerg Med 2011;18:215-20.



- 13. Lamantia MA, Stewart PW, Platts-Mills TF, et al. Predictive value of initial triage vital signs for critically ill older adults. West J Emerg Med 2013;14:453-460.
- 14. Cei M, Bartolomei C, Mumoli N. In-hospital mortality and morbidity of elderly medical patients can be predicted at admission by the Modified Early Warning Score: a prospective study. Int J Clin Pract 2009;63:591-5.
- 15. Modified Early Warning Score and VitalPac Early Warning Score in geriatric patients admitted to emergency department. Dundar ZD, Ergin M, Karamercan MA, Ayranci K, Colak T, Tuncar A, Cander B, Gul M. Eur J Emerg Med. 2016 Dec;23(6):406-412.
- 16. Epidemiological characteristics of geriatric patients in emergency departments: Results of a multicenter study. Ergin M, Karamercan MA, Ayranci M, Yavuz Y, Yavasi O, Serinken M, Acar T, Avcil M, Al B, Bayramoglu A, Durgun HM, Golcuk Y, Arziman İ, Dündar ZD. Turkish Journal of Geriatrics 2015; 18(4): 259-65

#### 3.2. Study objectives

#### MAIN OBJETIVE

The main objective of this project will be

- To determine Epidemiologic and Age Related Characteristics of Geriatric Patients presenting to the ED across Europe.

#### **SECONDARY OBJETIVES**

- To evaluate Early Warning Scoring systems (REMS, MEWS and VIEWS Scores) and determine most suitable Geriatric Emergency Medicine Risk Score regarding hospitalization, ICU admission and in-hospital mortality for patients
- To determine the most effective triage elements that can be used to predict hospitalization of geriatric patients presented to ED



- To determine the in hospital mortality and short term mortality rates of the patients above 65 years of age presenting to the ED across Europe.
- Sub analysis of ED discharged patients versus admitted patients for characteristics, comparison to recommended care and re-ED visit.
- Comparison of European data characteristics, investigation, treatment and outcome to similar data in other part of the world.

#### 4. STUDY DESIGN

#### 4.1. Study Design

Prospective non interventional cohort study in European EDs.

#### **5. SELECTION OF CASES**

#### 5.1. Setting

**Hospital Emergency Departments** 

#### **5.2. Population Selected**

Patients  $\geq$  65 years of age those presented to EDs with any symptom

#### 5.3. Inclusion criteria

- ✓ Consecutive geriatric patient presenting to the ED with any symptom
- ✓ 65 years or older

#### 5.3. Exclusion criteria

- ✓ No acceptance to participated
- ✓ End of life patients

#### 5.4. Variables included on the study

Variables are reflected on the Case Report Form



#### 5.5. Participation centres

Sites recruitment is still ongoing.

#### 5.6. Sample size

✓ All of the patients over 65 years who had presented to emergency services due to acute medical or surgical reasons during the 7 days study period are to be included. Patients younger than 65 years of age will be excluded from the study. The patients who had been brought to emergency services after having undergone cardio pulmonary resuscitation by the emergency medical team will be also excluded from the study.

 ✓ We strive for at least 25 patients per site per study period with a complete case report form (CRF). (This number is based on our pilot study, TEDGeS - Turkish Emergency Departments Geriatric Scoring Study)

✓ Each participating center will have to enroll all consecutive cases.

#### 5.7 Study period

7 consecutive days from 8:00 AM to 8:00 AM

#### 6. TREATMENT

No modification on the selected management is required.

#### 7. STUDY METHODOLOGY. INSTRUMENTS AND PROCEDURES

#### 7.1. Recruitment methodology.

Consecutive geriatric patient presenting to the ED during the selected study periods.

#### 7.2. Instruments

Case report form (CRF): Appendix 1



#### 8. ADVERS EVENTS

No intervention on establish management is requiring. Adverse events registry and declaration is no applicable.

#### 9. ETHICAL ASPÈCTS

#### 9.1. Ethical committees

Evaluation and acceptance of the protocol by local Ethical Committees is mandatory for each participating site.

#### 9.2. Inform consent

Depending the local regulation, an informed consent through a document might be needed.

#### 9.3. Confidentiality

No personal data is included on the database and all the CRF forms will be filled with 'CASTOR EDC' Clinical Data Management System, which enables secure data processes. Each center and country PI will be given a password to enter the data into CRF which will be secured and only be opened with the specific password or study managers' password.

#### 9.4. Good practices

Study should follow any local regulation related to good practices on medical research activities.

#### 10. LOGISTIC ASPECTS

#### 10.1. National Coordinator

There will be one national coordinator in each participating country. His responsibilities are:

- ✓ Select the participation centers.
- ✓ To be a link between the sites and the European PIs
- ✓ Participate on the final analysis and report.

#### 10.2. Case report form

Appendix 1



#### 10.3. Protocol

#### 10.3.1. Protocol modifications

Any change in the protocol has to be accepted by the EGERS steering committee and approved by the local ethics committee.

#### 10.3.2. Changes in the protocol during the recruitment period

No changes are accepted

#### 10.4. Data management

CRF are completed anonymously with 'CASTOR EDC' Clinical Data Management System, local researchers are responsible of quality in the information collected.

#### 10.4.1. Data collection

Promoter will provide the necessary tools (CRF) and online web access to transfer data into digital application to facilitated control and management and analysis.

#### 10.4.2. Data quality control

Specific indicators are establishing to evaluated quality of the information basically % of missing data for each variable and % on NA data on each variable.

#### 10.4.3. Data

Data bases will be collected and keep under control by the EGERS steering committee. Minimum time before deleting information is five years.

#### 10.5. Publications

Any publication has to refer to the original protocol and promoter EGERS EuSEM Research Network.

Any publication has to be communicated to National coordinators.

No use or transmission of data to a third party may be made without the prior consent of the EGERS Steering Committee

Each site will have access to its own data.

Each publication project must be submitted to the EGERS Steering Committee



#### 10.6. Data property

Data control and property belong to the promoter: EuSEM

#### 10.7. Author Ship

The EGERS Steering committee will be in charge of the coordination of all the articles that will be published.

The 1<sup>st</sup> author will be the one that writes the article

3 positions as authors will be dedicated to members of the EGERS Steering Committee

Position as author will also be dedicated to people who actually participated in the development of the protocol and in the drafting of the results and also the number of patients with a complete CRF.

#### 11. ANALYSIS

#### 11.1. Data Analysis

Patients will be classified based on their ages, emergency medicine diagnosis and early warning scores.

The normality analyses of the data will be performed using the Kolmogorov-Smirnov and Shapiro-Wilk tests. The data did not comply with normal distribution. The continuous variables will be expressed as the median (inter-quartile range), and the categorical variables were expressed as a number (percentage). The inter-group differences between the continuous variables will be evaluated using the Kruskal-Wallis test and the Mann-Whitney U test (with Bonferroni correction). The intergroup differences between the categorical variables will be evaluated using the Chi-square and Fischer Exact tests. The predictive power of the scores for hospitalization and mortality in hospital will be evaluated using the Receiver Operating Characteristic (ROC) analysis. The values of the Areas Under the ROC Curve (AUC) will be evaluated. The optimum cut-off points of the scores will be determined for both of the main endpoints using the Youden index (sensitivity+specificity-1).



Using these determined cut off points for the sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratio (+) and likelihood ratio (-), the values of both the scores will be calculated for both hospitalization and mortality at the hospital. Graph representation will be used to increase understanding of data.

#### 11.2. Missing data

Certain crucial variables are needed to accept a CRF as a useful one.

#### 11.3.1. Sample size

As this is a descriptive study, a formal sample size calculation has not been performed.

Based on our past experience of similar studies, we would expect to enroll between 40 and 50 sites each with an average number of patients of at least 25/site per 7 days study period.



**Appendix 1: Case Report Form** 

### **EGERS CRF**

# **European Geriatric Emergency Departments Registry Study**

| Inclusion criteria: All consecutive patients aged 65 or older presenting to the Emergency |
|---|
| Proposed study period, 7 consecutive days from 19th October 2020 to 16th November 2020: |
| First 3 Letters of the Country _ Site Patient N _ |
| Day of admission: Monday Tuesday Wednesday Thursday Fiday Saturday Sunday |
| Time of admission: \$\begin{aligned} 00:00-08 00 & \Boxed 08:01-16 00 & \Boxed 16:01-20 00 & \Boxed 20:01-23 59 \end{aligned}\$ |
| Gender: M F Age (yo) |



| Major Presenting Complaint: (Just Check One Major Complaint) | | | |
|---|---|---|---|
| Non-Traumatic Complaint | | Traumatic Complaint | |
| □ Abdominal Pain | | □ Falls | |
| <ul> <li>Agitation and Psychosis</li> </ul> | | | Motor Vehicle Accidents |
| | The Alcoholic Patient | | Pedestrian Struck |
| | Back Pain | | Burns |
| | Bleeding | | Assaults |
| | Chest Pain | | Other |
| | Dizziness (Vertigo) | | Trauma |
| | <b>Extremity Pain and Numbness</b> | | |
| | Fever (Elevated Temperature) | | |
| | Headache | | |
| | Hypotension | | |
| | Jaundice | | |
| | Mental Status Change and Coma | | |
| | Palpitations and Tachycardia | | |
| | Rash | | |
| | Seizure | | |
| | Shortness of Breath | | |
| | Syncope and Near-Syncope | | |
| | Toxic Ingestion | | |
| | Change in Vision | | |
| | Weakness and Fatigue | | |
| | Abnormal findings on examination of blood (Hyperglycemia, Anemia, etc) | | |
| | Other Non | | |
| | trauma | | |



| Presentation Symptoms and Signs: | | |
|---|---|---|
| Systolic Blood Pressure: _ mmHg | 7 | emperature: . ° C |
| Diastolic Blood Pressure: _ mmHg | F | Respiratory rate/min: _ |
| | Oxygen saturation (SpO2): % | |
| Heart Rate: _ bpm | | leeds additional oxygen supply with nasal cannula or ace mask: O Yes O No |
| Glasgow Coma Score: Eye: Voice: Moto | r: _ | _ TOTAL: |
| <u>Co-ma</u> | orb | idities: |
| Coronary artery disease | | Dyslipidemia Chronic |
| Left Ventricular Failure | | Liver disease |
| Right Ventricular Failure | | Chronic inflammatory disease |
| Prior coronary revascularization (Bypass) | | Active/recent malignant tumor |
| Chronic Obst. Pulm. Disease | | Anemia |
| Asthma | | Dementia, Alzheimer |
| Chronic renal disease wo routine dialysis | | Immunosuppression/AIDS |
| Chronic renal disease with routine dialysis | | Alcohol (> 30g/day for M and > 20 g/day for F) |
| Prior stroke (Hemorrhagic or Ischemic) | | Smoking (Active or stopped within last year) |
| Diabetes mellitus | | Other |
| Hypertension | | |
| Chron | ic I | Medications: |
| Beta-blockers | | Oral Antidiabetics |
| Calcium antagonists | | Insulin |
| ACE Inhibitors or Angiotensin II receptor | | Oral Steroids |
| blockers | | Cardiac Glycosides |
| Diuretics | | Vit K antagonists |
| Statins | | Psychiatric treatment |
| Antiplatelet | | Antidepressant |
| NSAID or Other Analgesics | | Antiepileptic |
| Inhaled Beta2mimetics | | Chemotherapy Drugs |
| Inhaled steroids | | Other |
| Oxygen +/- NIV at home | | |



| Consequence of ED Presentation: | |
|---|---|
| Final (Hospital or ED for discharged patients) Pr | incipal Diagnosis (only one diagnosis): |
| O Yes O No □ Patient Has History of Falls O Yes O No □ Patient Has Temporary Disorientation O Yes O No | For HOSPİTALİZED PATİENTS<br>STATUS at 30 days: |
| <ul> <li>□ Discharged From the Emergency Department Length of stay in ED:</li></ul> | If Admitted to Wards or ICU Total Length of Stay in Hospital: _ (days) Total Length of Stay in Wards: _ (days) Total Length of Stay in ICU: (days) Still in Wards Still in ICU |



# Appendix 2 **Country questionnaire** Number of ED proposed **Emergency Department Questionnaire** Institution: Address: **Local PI:** Last name: First name: Phone: e-mail address: How many patients per year do you receive in your Emergency Department (ED) How many patients per year do you hospitalize either in you hospital or in another hospital: Total number of patients presented to your ED during the study week Population served (habitants) by your ED Is your ED located in a: (check ONLY ONE BOX) General hospital: Teaching hospital: How many full time medical staff members do you have in your ED: How many full time nurse staff members do you have in your ED: No $\square$ Do you have an observation unit in your ED? Yes $\square$ Are patients admitted to the ED observation unit considered as hospitalized? Yes No Who perform the triage: Nurse Physician



| COMMITMENT TO CONFIDENTIALITY OF DATA |
|---|
| Dr./ Hospital |
| It is noted: |
| <ul> <li>To be undertaken the study entitled: "EGERS (European Geriatric Emergency Departments Registry Study)." by reviewing data from medical records, under the trial approved by the ethical Committee of research clinic of the Hospital</li> <li>Who undertakes to keep strict confidentiality of personal data from the source.</li> <li>Test results may be reported in congresses, meetings and scientific publications always safeguarding the confidentiality of personal data.</li> </ul> |
| Signature: Dr. |

In COUNTRY , DATE



#### PARTICIPANT INFORMED CONSENT PAPER

Research Project Title: EGERS (European Geriatric Emergency Departments Registry Study) Promoter: Dr./Dr.

I (name and surname of the patient or family member by specifying the degree)...

I have read the information sheet that it has given me.

I could do the study questions.

I have received sufficient information on the study.

I have spoken to: Dr/Dr. (name of the researcher)

I understand that my participation is voluntary.

I understand that I may withdraw my study:

- 1. Whenever
- 2. Without having to give explanations.
- 3. Without that this impact on my health care.

I freely provide my agreement to participate in the study.

| SIGNATURE of participant: | | |
|---------------------------|----|----|
| SIGNATURE of RESEARCHER | Dr | |
| | | ٠. |
| | | ٠. |
| DATE: | | |



#### **INFORMATION SHEET TO THE PATIENT**

The Study Title: EGERS (European Geriatric Emergency Departments Registry Study)
Promoter: Main RESEARCHER Mehmet Akif KARAMERCAN MD PhD, Chair of the
Geriatrics Special Interest Group of EuSEM Research Committee

#### INTRODUCTION

We are writing to inform you about a research study in which you are invited to participate. The study has been approved by the Committee of ethics of the research of the Hospital...., according to the legislation in force, and is carried out with respect for the principles contained in the Helsinki Declaration and the standards of good clinical practice. Our intention is just that you are receiving the correct information and sufficient so that you can evaluate and judge whether you want to or not to participate in this study. So read this fact sheet with attention and we will clarify any doubts that might arise after the explanation. In addition, you can consult with persons it deems appropriate.

VOLUNTARY PARTICIPATION: you should know that your participation in this study is voluntary and you can decide not to participate or change its decision and withdraw consent at any time, without therefore will alter the relationship with your doctor or causing prejudice in its treatment.

#### GENERAL DESCRIPTION OF THE STUDY:

The main objective of this project will be

- o To determine Epidemiologic and Age Related Characteristics of Geriatric Patients presenting to the ED across Europe.
- o To evaluate Early Warning Scoring systems and determine most suitable Geriatric Emergency Medicine Risk Score

#### **DESIGN OF THE STUDY:**

It is a prospective, observational, longitudinal, multicenter, multi-continental study. The estimated duration of study is three (3) months, will be carried out by the emergency room doctors of the emergency service of.... It does not involve risks for the patient.

Thanks to your cooperation in the present study, the population of the European Union, will benefit and therefore it may save lives, which would not be possible without their collaboration, and this study. There is no problem in the participation of women in fertile age. The treatment that will receive is not going to be changed by its involvement in the study. The doctor responsible for the study (Dr/Dra), can provide you more information, if desired.



Data collected for the study will be identified by a code and only your doctor's study and collaborators can relate this data with you and your medical history. Therefore, your identity will not be disclosed to any other person.

**COMPENSATION**: your participation in the study does not imply you any expenses.

**OTHER RELEVANT INFORMATION**: if you decide to withdraw the consent to participate in this study, no new data will be added to the database, and it may require the destruction of all identifiable samples previously retained to prevent the implementation of new analysis, while those responsible for the study may continue to use information collected about you until then, unless you expressly object. If you is removed from the study, by some of the expressed reasons, your doctor will prescribe a treatment appropriate to his illness. By signing the attached consent sheet, undertakes to comply with the procedures of the study explained him.

In COUNTRY, DATE

Dr.